CLINICAL TRIAL: NCT04127461
Title: Endoscopic Harvesting of the Radial Artery and Saphenous Vein Grafts in Coronary Artery Bypass Surgery.
Brief Title: Endoscopic Harvesting in Coronary Artery Bypass Grafting.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Gianluigi Bisleri (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor-Investigator, Dr. Gianluigi Bisleri, Associate Professor, Department of Surgery, Queen's University, Queen's University
Organization: Queen's University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: SURG-400-17
Record Dates: First submitted 2019-09-24; First posted 2019-10-15 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Coronary Bypass Stenosis; Graft Infection

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: retrospective data collection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Open vessel harvesting (Active Comparator): Arm 1 is the conventional procedure
  Interventions: Device: Medtronic endoscope
- Medtronic endoscope (Experimental): Arm 2 - is the minimally invasive procedure
  Interventions: Device: Medtronic endoscope

INTERVENTIONS:
Device: Medtronic endoscope — The endoscope is a minimally invasive tool used to remove veins from the leg traditionally used for CABG.

SUMMARY:
This is a retrospective data collection looking at patients who received either an endoscopic vessel harvesting procedure versus the conventional open procedure. Besides looking at cost variables in the 2 groups, other outcomes of interest include length of hospital stay, rates of infection, medication use, re-admissions and compilations.

DETAILED DESCRIPTION:
Since April 2018, the study database has been updated with all patients (currently there are 340 patients per group) and variables - both reflecting effectiveness of the procedure and cost. Preoperative variables being captured include comorbidity factors and variables relating to the Society of Thoracic Surgery (STS) score , which is a pre-procedure assessment of surgical risk.

The postoperative data collection includes a variety of complications and comorbidities the patient could experience during their hospital stay. These variables will provide us with information regarding procedure effectiveness, patient recovery and further costs associated with the procedure. Medications and antibiotics provided during the stay are also being captured. Total hospital costs will include any costs associated with ward stay, separated per level of care: Intensive Care Unit (ICU), Cardiac Surgical Unit (CSU), and regular ward.

The two follow up periods are 30 days and 6 months. Both look at the same effectiveness variables, any emergency room (ER) visits, re-admissions, and their respective reasons. Quality of life will be obtained by looking at the number of complications the patient experienced during these periods. The frequency of home care services provided to each patient, if any, are also being tracked. Cost calculations will be done by obtaining the time, length and number of visits to the ER, re-admissions and clinic visits.

ELIGIBILITY:
Inclusion Criteria:

* any patient at the KHSC undergoing a CABG procedure requiring a vein graft.

Exclusion Criteria:

* undergoing a simultaneous procedure.

Ages: 19 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 773 (Actual)
Dates: Start 2016-09-03 (Actual); Primary Completion 2018-12-20 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
cost analysis | 6 months
  economic cost of open versus endoscopic vessel harvesting

SECONDARY OUTCOMES:
Length of stay | 2 days
  days beyond normal length of stay
infection | 6 months
  infection of graft harvesting site